CLINICAL TRIAL: NCT00490165
Title: Associations Between Periodontal and Periapical Inflammation and Pregnancy Outcomes
Brief Title: Periodontal and Periapical Inflammation and Pregnancy
Status: Completed | Type: Observational
Sponsor: Roger Johnson (Other)
Responsible Party: Sponsor-Investigator, Roger Johnson, Professor, University of Mississippi Medical Center
Organization: University of Mississippi Medical Center (Other)
Other Study IDs: 2006-0198
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Periodontal Disease; Periapical Disease; Pregnancy; Diabetes; Cardiovascular Disease; Dental Caries
MeSH Terms: conditions — Periodontal Diseases; Periapical Diseases; Diabetes Mellitus; Cardiovascular Diseases; Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective chart review of patient records at the University of Mississippi Medical Center. We are not actively recruiting patients for this study. Recent animal studies we conducted showed that periapical abscesses during pregnancy cause a systemic inflammatory response in the mother. Also due to the increase in TNF-alpha (an inflammatory cytokine) the mother also become insulin resistant and thus developed gestational diabetes. Periodontal inflammation has been shown in the research to lead to low-birth weight and pre-term birth. We are looking retrospectively to see if an association exists in charted data between periapical and periodontal inflammation and adverse pregnancy outcomes.

DETAILED DESCRIPTION:
A. Specific Aims

1. To determine possible associations between periapical oral infection and adverse pregnancy outcomes in female patients in the School of Dentistry, the Dental/Dental Emergent Care Clinic (Jackson Medical Mall), and the UMC Hospital.
2. To examine the effects of several confounding variables related to stress from pain from the periapical infections on these adverse outcomes.

B. Background and Significance

During the past five years there has been increasing evidence for associations between periodontal infection and adverse pregnancy outcomes in humans, including preterm birth, low birth-weight babies, gestational diabetes, miscarriage, and preeclampsia. These events likely result from oral infections because bacteremia and release of pro-inflammatory cytokines from the diseased oral sites have been described.

Proinflammatory cytokines have been reported to be harmful and destructive to a successful pregnancy. The adverse fetal inflammatory response to TNF-alpha, IL-6 and C-reactive protein has been associated with preterm birth. These cytokines are also commonly associated with oral infections, both periodontal and periapical11. In addition, oral infections often produce pain and stress, which are considered harmful to a successful pregnancy. Since the effects of periodontal infections on adverse pregnancy outcomes have been described, it would be worthwhile to examine the specific effects of oral periapical abscesses on adverse birth outcomes, to begin to determine whether there is an association between this type of oral infection and these adverse outcomes.

There is no published information concerning the possible associations of tooth abscesses on pregnancy outcomes. In addition, there is no known biological mechanism for the direct link between periodontal infections, pre-term birth and low birth-weight babies. Secondary factors such as age, race, and life-style likely confound assessment of these associations. There are some preliminary studies of these variables in regard to the association between periodontal infections and adverse pregnancy outcomes, but not for periapical lesions. Since periapical lesions produce pain, these secondary factors could be more important to pregnancy outcomes than the primary factors (bacteria and proinflammatory cytokines).

C. Data collection. Archived dental records from female patients treated during the past three years at the University of Mississippi School of Dentistry and the Dental/Dental Emergent Care Clinic (Jackson Medical Mall) will be examined. Each patient record will be assigned a study number, and data will be entered on an Excel spreadsheet using that study number. Since the pregnancy outcome is part of the UMC Hospital record, the principal investigator will link the dental and hospital records using the patient name. However, the data collected will use a research number. Following the procedure for linking the patient records, the patient name will be discarded. Thus, it will not be possible to link an individual patient to the study data.

The following information will be recorded: age, pregnancy status, number of pulpal abscesses, number of sites of periodontitis (pocket depth ≥ 4 mm), race, highest level of education, DMFT (decayed, missing, filled teeth), number of children, past pregnancy outcomes, diagnosis of diabetes mellitus, and any other known pregnancy related conditions experienced during previous pregnancies from the records of the Dental/Emergent Dental Care Clinic. We will define adverse pregnancy outcomes as gestational diabetes, preeclampsia, pre-term birth, and a low-birthweight infant from the UMC hospital records.

D. Statistical Analysis of data. The data will be analyzed using SPSS v12 using appropriate statistical tests, including factorial ANOVA with post hoc tests, multivariate logistic regression, the Spearman correlation test, and chi square analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Child bearing age or above

Exclusion Criteria:

* Male
* Very young children (before child-bearing age)

Min Age: 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We are looking at charts of patients (former patients) at the University of Mississippi School of Dentistry. Since this is a pregnancy study we are looking only at the charts of female patients. The youngest record we review is 10 and there is no upper limit to the age.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Bain, BS, Principal Investigator — University of Mississippi Medical Center; Roger Johnson, PhD; DMD, Study Director — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States